CLINICAL TRIAL: NCT05061342
Title: Tumor Control, Treatment Toxicity, Quality of Life and Bio-Imaging Repository Databank (TQ-BIRD) for Cancer Patients-A Master Protocol for Imaging and Blood Biomarker Group
Brief Title: Tumor Control, Treatment Toxicity, Quality of Life and Bio-Imaging Repository Databank (TQ-BIRD) for Cancer Patients
Acronym: TQ-BIRD
Status: Recruiting | Type: Observational
Sponsor: Fengming Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Taizhou Hospital (Other); Peking University Shenzhen Hospital (Other); Shenzhen People's Hospital (Other); The First Affiliated Hospital of Henan Medical University (Unknown)
Responsible Party: Sponsor-Investigator, Fengming Kong, Tenured Clinical Professor, The University of Hong Kong-Shenzhen Hospital
Organization: The University of Hong Kong-Shenzhen Hospital (Other)
Other Study IDs: GCOG0001
Record Dates: First submitted 2021-05-21; First posted 2021-09-29 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: surgery; systemic therapy; radiotherapy; biomarker; imaging; toxicity; quality of life
MeSH Terms: conditions — Neoplasms | interventions — Observation; Radiotherapy; Medicine, Chinese Traditional; Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood, tissue, feces and body fluids such as urine, saliva, pleural effusion, ascites, and cranial spinal fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer Patients: Those with cancer.
  Interventions: Other: No experimental interventions 1. Observation; 2. Anticancer treatments, including surgery, systemic therapy, radiotherapy, Chinese traditional medicine, or palliative/supportive care.
- Normal (non cancer) controls: Those without cancer.

INTERVENTIONS:
Other: No experimental interventions 1. Observation; 2. Anticancer treatments, including surgery, systemic therapy, radiotherapy, Chinese traditional medicine, or palliative/supportive care. — Any anticancer or palliative care
  Other Names: 1. Observation; 2. Anticancer treatments, including surgery, systemic therapy, radiotherapy, Chinese traditional medicine, or palliative/supportive care.
  Groups: Cancer Patients

SUMMARY:
Our central hypothesis is that patient response to treatment, evaluated by full spectrum of outcome measures including tumor control, survival, toxicity, and quality of life (QoL), will correlate with biomarker expressions, which can be tested in the blood, other body fluid, imaging as well as tumor tissue (if available).

DETAILED DESCRIPTION:
The primary biomarkers of our interest are those obtained from minimally invasive procedures and those associated with immune/inflammatory treatment responses such as lymphocyte count, immune cell subtype distribution, TGF-beta1, immunomodulating interleukins and IDO metabolites. We will measure the biomarkers pre-, during- and post-anticancer treatment for hypothesis driven studies, and bank residual biological specimen, in combination with prospectively collected data including patient/tumor/treatment factors, imaging, tumor control outcome, treatment toxicity and QOL measures. We will classify the tumor response according to RECIST criteria and qualify QoL by using the PROMIS grading system and correlate them with the corresponding biomarkers. This study will serve young investigators who are interested in biomarker studies for early diagnosis, tumor control outcome and treatment toxicity/QOL prediction, aiming to guide personalized cancer care in future.

ELIGIBILITY:
Inclusion Criteria:

Cancer Patients

* 18 years of age and older.
* Scheduled to receive any kind of therapy in our center.
* Performance status of ECOG 0, 1, 2, or 3.
* Able to understand QoL questionnaire.

Normal (non cancer) controls

* 18 years of age and older healthy volunteers.
* Without a history of cancer except for cured skin cancer, without any active cancer.
* ECOG Performance status 0, 1, 2, or 3.

Exclusion Criteria:

Participants who have supposedly limited ability to complete the survey questionnaires of the present study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients received any form of treatment (radiotherapy, surgery, systemic therapy, palliative and alternative cares) in the cancer center will be invited to participate. Patients with clinical diagnosis of tumor or related diseases such as hepatitis, gastritis, and Myasthenia Gravis will also be eligible, particularly should the patient be taken to OR for such treatments or being monitored for the risk of cancer developments. Healthy volunteers of various ages will also be enrolled from the general public for controls and setting up normal ranges of the interested biomarkers.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor control, treatment toxicity, quality of life | Changes of treatment toxicity and quality of life will be evaluated before, during and after treatment until 2 years after treatment. Treatment efficacy including tumor control will be evaluated until patients' death or lost to follow-up.
  Changes of treatment-related adverse events as assessed by CTCAE v5.0, and changes of quality of life as assessed by PROMIS-29 Profile v2.1. from baseline, during and after treatment until 2 years after treatment.
  Tumor response, tumor control, progression-free survival (PFS), cause-specific survival (CSS) and overall survival (OS) evaluated until patients' death or lost to follow-up.
  Changes of treatment-related adverse events as assessed by CTCAE v5.0, and changes of quality of life as assessed by PROMIS-29 Profile v2.1. from baseline, during and after treatment until 2 years after treatment. Tumor response, tumor control, progression-free survival (PFS), cause-specific survival (CSS) and overall survival (OS) evaluated until patients' death or lost to follow-up.

SECONDARY OUTCOMES:
Bio-Imaging-Repository-Databank (BIRD) | Blood, feces, urine and saliva will be collected, whenever possible before, during and after treatment for at least four times (baseline, middle, at the end and the first follow-up around 1-3 months after treatment.
  Prospectively collect and store body fluids samples from cancer patients treated with various anticancer treatments, including palliative care to establish a bio-Imaging-repository-databank covering an extensive repository and prospective clinically relevant data.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ming (Spring) KONG, Professor, Principal Investigator — The University of Hong Kong-Shenzhen Hospital
Locations (1):
- UHongKongShenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao CN, Chiang CL, Chiu WK, Chan SK, Li CJ, Chen WW, Zheng DY, Chen WQ, Ji R, Lo CM, Jabbour SK, Chan CA, Kong FS. Treatments of transarterial chemoembolization (TACE), stereotactic body radiotherapy (SBRT) and immunotherapy reshape the systemic tumor immune environment (STIE) in patients with unresectable hepatocellular carcinoma. J Natl Cancer Cent. 2024 Nov 28;5(1):38-49. doi: 10.1016/j.jncc.2024.06.007. eCollection 2025 Feb. PMID 40040869